CLINICAL TRIAL: NCT03520205
Title: Comparison Between Quadratus Lumborum Block and Epidural on Stress Response and Perioperative Cellular Immunological Function of Laparoscopic Nephrectomy Kidney Donor
Brief Title: Quadratus Lumborum Block Versus Epidural for Laparoscopic Nephrectomy Kidney Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes021
Record Dates: First submitted 2018-04-15; First posted 2018-05-09 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Renal Transplant Donor of Left Kidney
Keywords: stress response; kidney donor; Cellular Imunological Function; quadratus lumborum block; numerical rating scale; morphine patient controlled analgesia
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Active Comparator): Patient will receive quadratus lumborum block
  Interventions: Procedure: Quadratus Lumborum Block
- Continuous Epidural (Active Comparator): Patient will receive epidural anesthesia
  Interventions: Procedure: Continuous Epidural

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Bilateral block using ultrasound will be performed before surgery and after surgery on patient using Stimuplex 100mm needle with Bupivacaine 0.25% 0.4 mL/kg, maximum dose 25 mL each side under general anaesthesia
  Arms: Quadratus Lumborum Block
Procedure: Continuous Epidural — Patient will be given 6 mL/hour of Bupivacaine 0.25% for intraoperative analgesia and continued epidural 6 mL/hour Bupivacaine 0,125% as postoperative analgesia in 24 hours.
  Arms: Continuous Epidural

SUMMARY:
This study aimed to compare Quadratus Lumborum Block to Epidural on Stress Response and Perioperative Cellular Immunological Function of Laparoscopic Nephrectomy Kidney Donor

DETAILED DESCRIPTION:
Sixty-two subjects were given informed consent before enrolling the study and randomized into two groups; quadratus lumborum block and epidural. Non-invasive blood pressure monitor, electrocardiogram (ECG), and pulse-oxymetry were set on the subjects in the operation room. General anesthesia induction was done by fentanyl 2 mcg/kg and propofol 1-2 mg/kg. Endotracheal tube (ETT) intubation was facilitated with Atracurium 0.5mg/kg as muscle relaxant. Maintenance was done by sevoflurane, oxygen, and compressed air. On quadratus lumborum block group, bilateral block using ultrasound will be performed with stimuplex 100mm needle with 20 cc of bupivacaine 0.25% as regimen. On epidural group, epidural catheter was inserted under general anaesthesia on left lateral decubitus position (5 cm depth inside the epidural space) at level Th10-Th11. The catheter insertion was confirmed with vacuum aspiration and negative test-dose. Before first incision, patient will be given continuous epidural Bupivacaine 0.25% 6 mL/hour. Blood sample was drawn for interleukin-6, blood glucose, and c-reactive protein as baseline data. After surgery, patient were extubated until fully conscious and can follow command verbally. Patient will be transported in recovery room post operation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney donor patients undergoing laparoscopic nephrectomy
* Body mass index below 30
* Duration of surgery 4 to 6 hours
* Patients who agreed to participate in this study and sign informed consent.

Exclusion Criteria:

Have contraindication for quadratus lumborum block

* Have contraindication for epidural
* Previous history of local anesthetic drug allergy
* inability to communicate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Interleukin-6 at 24 hours after abdominal insufflation | Before procedure, at the end of surgery, and 24 hours after abdominal insufflation
  Measure by ELISA
Cumulative morphine requirement at 2 hours, 6 hours, 12 hours, 24 hours postoperative | 2 hours, 6 hours, 12 hours, 24 hours.
  Cumulative morphine consumption at each time point in 24 hours after surgery

SECONDARY OUTCOMES:
Change from Baseline Patient Controlled Analgesia at 2, 6, 12 and 24 hours after procedure | 2, 6, 12, and 24 hours after procedure
  Measure by how many times patient use morphine PCA analgesia
Change from Baseline Pain Intensity at 2, 6, 12, and 24 hours after procedure | 2, 6, 12, and 24 hours after procedure
  Measured by Numerical Rating Scale
Change from Baseline Blood Glucose at 2 hours after abdominal insufflation | Before procedure and 2 hours after abdominal insufflation
  Measured by finger-stick blood sample
Change from Baseline Blood pressure | Intraoperative and 24 hours
  Measured by non-invasive blood pressure monitoring at before anaesthesia induction (baseline), post-induction, gas-insufflation, Pfannenstiel incision, end of surgery, and 24 hours surgery
Change from Baseline Mean Arterial Pressure | Intraoperative and 24 hours
  Measured by non-invasive blood pressure monitoring at before anaesthesia induction (baseline), post-induction, gas-insufflation, Pfannenstiel incision, end of surgery, and 24 hours surgery
Change from Baseline Cardiac Index | Intraoperative and 24 hours
  Measured by cardiometry ICON® at before anaesthesia induction (baseline), post-induction, gas-insufflation, Pfannenstiel incision, end of surgery, and 24 hours surgery
Change from Baseline Heart Rate | Intraoperative and 24 hours
  Measured by pulse oximetry at before anaesthesia induction (baseline), post-induction, gas-insufflation, Pfannenstiel incision, end of surgery, and 24 hours surgery
Change from Baseline hs-CRP at 48 hours after abdominal insufflation | Before procedure, at the end of surgery, and 48 hours after abdominal insufflation
  Measured with ELISA
Time to first morphine requirement | 24 hours
  Duration from end of anesthesia until first attempt of morphine requirement in minutes
Total bupivacaine used in 24 hours | 24 hours
  Total bupivacaine used until 24 hours postoperatively
Change from baseline motor block at 2, 6, 12, and 24 hours after anesthesia recovery | 2, 6, 12, and 24 hours after procedure
  Measured by Bromage score
Number of participants with paresthesia after procedure | 24 hours
  in percentage
Duration of urinary catheter | 24 hours
  in hours
Level of sensory block after procedure | 24 hours
  Measured by cold and pin prick sensation

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] SarinKapoor H, Kaur R, Kaur H. Anaesthesia for renal transplant surgery. Acta Anaesthesiol Scand. 2007 Nov;51(10):1354-67. doi: 10.1111/j.1399-6576.2007.01447.x. PMID 17944639
- [Background] Minnee RC, Idu MM. Laparoscopic donor nephrectomy. Neth J Med. 2010 May;68(5):199-206. PMID 20508268
- [Background] Buunen M, Gholghesaei M, Veldkamp R, Meijer DW, Bonjer HJ, Bouvy ND. Stress response to laparoscopic surgery: a review. Surg Endosc. 2004 Jul;18(7):1022-8. doi: 10.1007/s00464-003-9169-7. Epub 2004 May 12. PMID 15136930
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Das W, Bhattacharya S, Ghosh S, Saha S, Mallik S, Pal S. Comparison between general anesthesia and spinal anesthesia in attenuation of stress response in laparoscopic cholecystectomy: A randomized prospective trial. Saudi J Anaesth. 2015 Apr-Jun;9(2):184-8. doi: 10.4103/1658-354X.152881. PMID 25829908
- [Background] Gulyam Kuruba SM, Mukhtar K, Singh SK. A randomised controlled trial of ultrasound-guided transversus abdominis plane block for renal transplantation. Anaesthesia. 2014 Nov;69(11):1222-6. doi: 10.1111/anae.12704. Epub 2014 Jun 28. PMID 24974901
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Skrekas G, Papalois VE, Mitsis M, Hakim NS. Laparoscopic live donor nephrectomy: a step forward in kidney transplantation? JSLS. 2003 Jul-Sep;7(3):197-206. PMID 14558706
- [Background] Oyen O, Scholz T, Hartmann A, Pfeffer P. Minimally invasive kidney transplantation: the first experience. Transplant Proc. 2006 Nov;38(9):2798-802. doi: 10.1016/j.transproceed.2006.08.102. PMID 17112833
- [Background] Jianda X, Yuxing Q, Yi G, Hong Z, Libo P, Jianning Z. Impact of Preemptive Analgesia on inflammatory responses and Rehabilitation after Primary Total Knee Arthroplasty: A Controlled Clinical Study. Sci Rep. 2016 Aug 31;6:30354. doi: 10.1038/srep30354. PMID 27578313
- [Background] Southworth SR, Woodward EJ, Peng A, Rock AD. An integrated safety analysis of intravenous ibuprofen (Caldolor((R))) in adults. J Pain Res. 2015 Oct 23;8:753-65. doi: 10.2147/JPR.S93547. eCollection 2015. PMID 26604816
- [Background] Spiro MD, Eilers H. Intraoperative care of the transplant patient. Anesthesiol Clin. 2013 Dec;31(4):705-21. doi: 10.1016/j.anclin.2013.09.005. Epub 2013 Nov 6. PMID 24287348
- [Background] Bhosale G, Shah V. Combined spinal-epidural anesthesia for renal transplantation. Transplant Proc. 2008 May;40(4):1122-4. doi: 10.1016/j.transproceed.2008.03.027. PMID 18555130
- [Derived] Aditianingsih D, Pryambodho, Anasy N, Tantri AR, Mochtar CA. A randomized controlled trial on analgesic effect of repeated Quadratus Lumborum block versus continuous epidural analgesia following laparoscopic nephrectomy. BMC Anesthesiol. 2019 Dec 5;19(1):221. doi: 10.1186/s12871-019-0891-7. PMID 31805855
- See also: STRESS RESPONSE AND ANAESTHESIA ALTERING THE PERI AND POST-OPERATIVE MANAGEMENT — http://medind.nic.in/iad/t03/i6/iadt03i6p427.pdf
- See also: Efficacy of parecoxib on the level of IL-6, CRP, and postoperative pain relief after percutaneous nephrolithotomy — http://www.ijcem.com/files/ijcem0028816.pdf